CLINICAL TRIAL: NCT06632236
Title: 5G-EMERALD: A Phase 1 Trial of Amivantamab in High Grade Malignant Brain Tumours Within the 5G Platform
Brief Title: 5G-EMERALD: Amivantamab in Malignant Brain Tumours
Acronym: 5G-EMERALD
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Institute of Cancer Research, United Kingdom (Other)
Collaborators: Royal Marsden NHS Foundation Trust (Other); Cambridge University Hospitals NHS Foundation Trust (Other); Janssen Pharmaceutica N.V., Belgium (Industry); Cancer Research UK (Other); Minderoo Foundation (Unknown); University of Cambridge (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: CCR5880
Record Dates: First submitted 2024-10-02; First posted 2024-10-09 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Malignant Primary Gliomas; Glioblastoma Multiform (Grade IV Astrocytoma); Diffuse Hemispheric Glioma, H3 G34-Mutant; Glioblastoma Multiforme (GBM)
MeSH Terms: conditions — Glioblastoma | interventions — amivantamab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experimental: Phase 1b (Experimental): The Phase 1b will evaluate the safety and tolerability of amivantamab and determine its preliminary antitumour activity when administered at the recommended Phase 2 dose (RP2D) in patients with molecularly defined malignant brain tumours.
  Interventions: Drug: Amivantamab

INTERVENTIONS:
Drug: Amivantamab — Amivantamab will be supplied in single-use 350 mg injectable solution, provided as a 7 ml per glass vial (50mg/ml), intended for IV infusion.
  Other Names: JNJ-61186372

SUMMARY:
The purpose of this clinical trial is to evaluate the safety and tolerability of amivantamab and to determine the preliminary antitumour activity of amivantamab administered at the recommended Phase 2 dose (RP2D). In the Phase 1b of this study a biomarker defined arm will be opened, initially in the relapsed GMB setting, enrolling 12 patients. These patients will be treated with amivantamab monotherapy. Amivantamab will be administered intravenously (IV) weekly for the first 4 weeks, then every 2 weeks thereafter until disease progression or unacceptable toxicity. The first dose will be given as a split infusion, 350 mg IV over 4 hours on cycle 1 day 1 and 1400 mg IV over 6 hours on cycle 1 day 2. Subsequent infusions are given at a dose of 1750 mg IV over 2-5 hours in cycle 1 and between 2-3 hours from cycle 2 onwards if the first dose was well-tolerated with no significant toxicity.

Progression to Phase 2 is dependent on emergent data and funding.

DETAILED DESCRIPTION:
The clinical trial will start in Phase 1b (proof of concept of hypothesis-driven biomarker-guided therapies).

This is a study within Minderoo 5G: A Next Generation AGile Genomically Guided Glioma Modular Platform for proof-of-concept molecular hypothesis testing in patients with high grade malignant brain tumours.

5G-EMERALD is a Bayesian multi-centre, multi-arm, open-label, adaptive, seamless Phase 1 trial of amivantamab for patients with high grade malignant brain tumours.

5G-EMERALD will recruit patients with glioblastoma (GBM) into one molecularly-defined biomarker arm of patients who have tumours that harbour:

• EGFR amplification (high copy number)

The above mentioned arm, within Phase 1, will have robust GO/ADAPT decision points, reviewed by the Safety Review Committee (SRC) to allow for both agility and clear direction for next steps. A 2-stage Bayesian adaptive design will be performed to assess preliminary efficacy.

In the Phase 1b of this study a biomarker defined arm will be opened, initially in the relapsed GBM setting, enrolling 12 patients onto each arm. These patients will be treated with amivantamab. Amivantamab will be administered intravenously (IV) weekly for the first 4 weeks, then every 2 weeks thereafter until disease progression or unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria for Phase 1b:

1. Patients with histologically confirmed advanced WHO Stage IV glioblastoma (per fourth edition 2016). Per the new 2021 fifth edition of WHO Classification of Tumours of the Central Nervous System, this will include:

   * Glioblastoma, IDH-wildtype Grade 4
   * Astrocytoma, IDH-mutant, Grade 4 (lower Grade 2/3 are not included)
   * Diffuse hemispheric glioma, H3 G34 mutant Grade 4
2. Patients for Phase 1 will need to have consented to the Minderoo Precision Brain Tumour Programme and have available whole genome, and transcriptome data available.
3. Patients for the relapsed cohorts will be eligible at first relapse following completion of optimal surgery, and Stupp based adjuvant chemo-radiotherapy (or equivalent). They will need to have measurable disease per Response Assessment in Neuro-Oncology (RANO) or evaluable disease.
4. Patients for the front line minimal residual disease (MRD) cohort will be eligible following completion of optimal surgery and Stupp based adjuvant chemoradiotherapy as long as they meet all other inclusion/exclusion criteria.
5. 16 years or over.
6. Life expectancy of at least 12 weeks.
7. World Health Organisation (WHO) performance status of 0-1.
8. Neurologically stable (e.g., without a progression of neurological symptoms or requiring escalating doses of systemic steroid therapy within the last week).
9. Written (signed or dated) informed consent and be capable of co-operating with treatment and follow up.
10. Haematological and biochemical indices within the ranges shown below. These measurements must be performed within one week prior to the first dose of either IMP:

    Haemoglobin (Hb): ≥ 10.0 g/dL Absolute neutrophil count: ≥ 1.5 x 10^9/L Platelet count: ≥ 75 x 10^9/L Coagulation: INR <1.5 and APTT <1.5x if not anticoagulated INR stable > 7 days within intended therapeutic range if anticoagulated Bilirubin: ≤ 1.5 x ULN; subjects with Gilbert's syndrome can enrol if conjugated bilirubin is within normal limits.

    Alanine aminotransferase (ALT) and aspartate aminotransferase (AST): < 3 x ULN Albumin: ≥ 28 g/L Creatinine: <1.5 x ULN and creatinine clearance > 45 ml/min as measured or calculated based on Cockcroft-Gault formula Sodium: ≥ 130 mmol/L Potassium, Calcium, Magnesium, phosphate: Within institution normal ranges (replacement is permitted) Urinary protein: < 1+ on dipstick
11. Female patients with reproductive potential must have a negative serum, or urine, pregnancy test at screening and within 72 hours of the first dose of study treatment and must agree to further serum or urine pregnancy tests during the study.
12. A participant must be either of the following: a. not of childbearing potential, b. of child-bearing potential and practicing true abstinence during the entire period of the study, including up to 6 months after the last dose of the study treatment is given, or c. of childbearing potential and practicing 2 methods of contraception, including 1 highly effective user independent method and a second method, to avoid impregnating a partner or becoming pregnant, respectively. A participant must agree to continue contraception throughout the study, and for at least 6 months after the last dose of study treatment.

    Please, refer to section 4.1 of CTFG guidance "Recommendations related to contraception and pregnancy testing in clinical trials" and to section 9.6 of the Master Protocol for further details.

    Note: If the childbearing potential changes after start of the study (eg, participant of childbearing potential who is not heterosexually active becomes active, premenarchal participant experiences menarche) the participant must begin birth control, as described above.
13. A participant must agree not to donate eggs (ova, oocytes) for the purposes of assisted reproduction during the study and for 6 months after receiving the last dose of study treatment.
14. A participant must wear a condom when engaging in any activity that allows for passage of ejaculate to another person during the study and for 6 months after receiving the last dose of study treatment. A participant who is sexually active with a partner of childbearing potential must agree to use a condom with spermicidal foam/gel/film/cream/suppository and their partner must also be practicing a highly effective method of contraception (ie, established use of oral, injected, or implanted hormonal methods of contraception; placement of an intrauterine device [IUD] or intrauterine hormone-releasing system [IUS]). If the participant is vasectomized, they must still use a condom (with or without spermicide) for prevention of passage of exposure through ejaculation, but their partner is not required to use contraception.
15. A participant must agree not to donate sperm for the purpose of reproduction during the study and for a minimum of 6 months after receiving the last dose of study treatment.
16. A participant must be willing and able to adhere to the lifestyle restrictions specified in this protocol.

Exclusion Criteria for Phase 1b:

1. Receipt of treatment before the first dose of study drug (Cycle 1 Day 1) within an interval shorter than the following, as applicable:

   * Cytotoxic chemotherapy during the prior 2 weeks or 6 weeks for nitrosoureas
   * Bevacizumab during the prior 6 weeks
   * Five half-lives of any small molecule investigational or licensed medicinal product.
2. Prior immune checkpoint inhibitor therapy or vaccine therapy is not permitted. Prior EGFR-targeting therapy is not permitted. Prior use of any other immune-modulatory investigational agent must be discussed with sponsor team and CI.
3. Ongoing Grade 2 or greater toxicities from pre-existing conditions or from previous treatments.
4. Patients with carcinomatous meningitis, leptomeningeal spread of tumour, spread of tumour to the brain stem or spinal cord.
5. Has evidence of recent intratumoural or peritumoural haemorrhage on baseline MRI. Patients with radiological findings that are stable on at least 2 consecutive MRI scans at least 3 weeks apart will be eligible.
6. History of clinically relevant bleeding disorders, including significant gastrointestinal (GI) bleeding within last 6 months.
7. Participant has active cardiovascular disease including, but not limited to:

   * A medical history of deep venous thrombosis or pulmonary embolism within 1 month prior to first dose of study drug or any of the following within 6 months prior to first dose of study drug: myocardial infarction, unstable angina, stroke, transient ischemic attack, coronary/peripheral artery bypass graft, or any acute coronary syndrome. Clinically non-significant thrombosis such as non-obstructive catheter-associated thrombus, incidental or asymptomatic pulmonary embolism, are not exclusionary. Patients on Warfarin will need to be converted onto low-molecular weight-based heparin therapy.
   * Participant has a significant genetic predisposition to venous thromboembolic (VTE) events such as Factor V Leiden.
   * Participant has a prior history of VTE and is not on appropriate therapeutic anticoagulation as per National Comprehensive Cancer Network (NCCN) or local guidelines.
   * Uncontrolled (persistent) hypertension: systolic blood pressure > 160 mm Hg; diastolic blood pressure > 100 mm Hg.
   * Congestive heart failure (CHF), defined as New York Heart Association (NYHA) class III-IV or hospitalization for CHF (any NYHA class) within 6 months of first dose of the study drug.
   * Concurrent and clinically significant abnormalities on ECG at Screening, including a corrected QT interval (QTcF > 460ms).
8. History of malabsorption syndrome or other conditions that may interfere with enteral absorption. Patients with a history of or active inflammatory bowel disease (e.g., Crohn's disease or ulcerative colitis). Patients with acute or chronic pancreatitis. History of GI perforation or fistulae.
9. Has urine protein > 1g/24 hours. Participants with > 1+ on urine dipstick testing will undergo 24-hour urine collection for quantitative assessment of proteinuria.
10. Has significant lung disease including pneumonitis, interstitial lung disease (including drug-induced or radiation ILD/pneumonitis), idiopathic pulmonary fibrosis, cystic fibrosis, active tuberculosis, or history of opportunistic infections (including PCP or Cytomegalovirus (CMV) pneumonia).
11. Participant is serologically positive for hepatitis B surface antigen (HbsAg), Note: participants with a prior history of hepatitis B virus (HBV) demonstrated by positive hepatitis B core antibody are eligible if they have at Screening 1) a negative HBsAg and 2) a HBV DNA (viral load) below the lower limit of quantification, per local testing. Subjects with a positive HBsAg due to recent vaccination are eligible if HBV DNA (viral load) is below the lower limit of quantification, per local testing.
12. Participant is serologically positive for hepatitis C antibody. Note: participants with a prior history of hepatitis C virus (HCV), who have completed antiviral treatment and have subsequently documented HCV RNA below the lower limit of quantification per local testing are eligible.
13. Participant has other clinically active infectious liver disease.
14. Participant is positive for human immunodeficiency virus (HIV), with 1 or more of the following:

    * Receiving antiretroviral therapy (ART) that may interfere with study treatment (consult sponsor for review of medication prior to enrolment).
    * CD4 count < 350 at screening
    * AIDS-defining opportunistic infection within 6 months of start of screening
    * Not agreeing to start ART and be on ART > 4 weeks plus having HIV viral load < 400 copies/mL at end of 4-week period (to ensure ART is tolerated and HIV controlled).
15. Participant has an uncontrolled illness, including but not limited to:

    * Uncontrolled diabetes
    * Ongoing or active infection (includes infection requiring treatment with antimicrobial therapy [participants will be required to complete antibiotics 1 week prior to starting study treatment] or diagnosed or suspected viral infection.
    * active bleeding diathesis
    * Impaired oxygenation requiring continuous oxygen supplementation
    * Psychiatric illness, social situation, or any other circumstances that would limit compliance with study requirements
    * Any ophthalmologic condition that is clinically unstable
16. Steroid requirement for neurological symptom control of > 3mg Dexamethasone per day (patients will allowed to enrol if they have been on a stable dose of steroids of equivalent or less than 3mg Dexamethasone for at least 5 days prior to Day 1 of Cycle 1).
17. Has received a live vaccine within 30 days of planned start of study therapy. Note: inactive vaccines including COVID vaccines are allowed prior to 1 week of Day 1 of Cycle 1).
18. Concurrent or prior malignancy other than the disease under study. The following exceptions require consultation with the Chief Investigator:

    1. Non-muscle invasive bladder cancer (NMIBC) treated within the last 24 months that is considered completely cured.
    2. Skin cancer (non-melanoma or melanoma) treated within the last 24 months that is completely cured.
    3. Non-invasive cervical cancer treated within the last 24 months that is considered completely cured.
19. Is a participant or plans to participate on another interventional clinical trial while taking part in this Phase 1 study. Participation in an observational trial would be acceptable.
20. A participant has major surgery excluding placement of vascular access or tumour biopsy, or had significant traumatic injury within 4 weeks before first dose of study drug or minor surgery within 2 weeks, or will not have fully recovered from surgery, or has surgery planned during the time the participant is expected to participate in the study. Note: Participants with planned surgical procedures to be conducted under local anaesthesia may participate.
21. A participant has palliative radiotherapy within 1 week of the firs dose of study drug,
22. Any other condition which in the investigator's opinion would not make the patient a good candidate for the clinical trial.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2024-10-09 (Actual); Primary Completion 2026-03-05 (Estimated); Study Completion 2027-03-05 (Estimated)

PRIMARY OUTCOMES:
Phase 1b - To evaluate the safety and tolerability of investigational agent in patients with malignant brain tumours | 18 months
  To identify the incidence, nature and severity of adverse events and laboratory abnormalities, with severity determined according to NCI CTCAE v5.0
Phase 1b - To determine the preliminary antitumour activity of the investigational agent administered at the RP2D in patients with molecularly defined malignant brain tumours | 18 months
  Antitumour activity will be defined on the basis of the following outcomes. If any of the following occur, patients will be considered to have clinically benefitted: For relapsed GBM: Achievement of overall response of CR or PR per Response Assessment in Neuro-Oncology (RANO) within 6 months or Free of disease progression or death at 6 months For front line unmethylated GBM (MRD): • Progression-free survival (PFS)

SECONDARY OUTCOMES:
Phase 1b - To identify molecular determinants of response and antitumour activity of the investigational agent in patients with molecularly selected brain tumours | 18 months
  Determination of biomarkers of response, including but not limited to changes in genomic, transcriptomic or immunological signatures from responders and non-responders using tumour sequencing analysis.

OTHER OUTCOMES:
Exploratory objective - To determine mechanisms of resistance to the investigational agent in patients with malignant brain tumours | 18 months
  Correlate antitumour activity of the investigational agent with the detection of putative predictive biomarkers of response and resistance in archival tumours, patient derived cells lines and plasma samples banked as part of the Minderoo Precision Brain Tumour Programme.
Exploratory objective - To assess putative predictive biomarkers of the investigational agent in patients with malignant brain tumours | 18 months
  Correlate treatment response with co-segregating mutational landscapes and identify mechanism of precision drug resistance e.g., on target vs off target, on pathway.
Exploratory objective - To identify putative precision therapy combinations with the potential for additive benefit | 18 months
  Plan rational combination therapies based on these results.

CONTACTS AND LOCATIONS:
Overall Officials: Juanita Lopez, MD, PhD, Study Director — National Health Service, UK
Locations (2):
- United Kingdom (2):
  - Cambridge University Hospitals, Cambridge
  - The Royal Marsden Hospital - Drug Development Unit, Sutton